CLINICAL TRIAL: NCT00842114
Title: Association of Rituximab to Immunochemotherapy With CVP + Interferon in Newly Diagnosed Follicular Lymphoma Patients With Intermediate-high FLIPI Score. Phase II Study.
Brief Title: Rituximab and CVP Plus Interferon for Follicular Non Hodgkins Lymphoma (NHL)
Acronym: LNH-Pro-05
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fundación Leucemia y Linfoma, Spain (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LNH-Pro-05; EudraCT Number:2005-004761-42
Record Dates: First submitted 2009-02-10; First posted 2009-02-12 (Estimated); Last update posted 2016-04-04 (Estimated); Status verified 2016-03

CONDITIONS: Non-Hodgkin's Lymphoma
Keywords: Intermediate-high FLIPI score; Follicular Lymphoma; Progression free survival
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, Follicular | interventions — Cyclophosphamide; Prednisone; Vincristine; MAX protein, human; Interferons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- R+CVP+IFN (Experimental): 8 cycles of Rituximab plus CVP chemotherapy (Bagley's et al) associated with Interferon for 12 weeks
  Interventions: Biological: R+CVP+IFN

INTERVENTIONS:
Biological: R+CVP+IFN — Immunochemotherapy
  Other Names: Mabthera -Rituximab (375 mg/sm, D1)/cycle; Cyclophosphamide (400 mg/sm, D 1-5)/cycle; Prednisone (100 mg/sm,D 1-5)/cycle; Vincristine (1.4 mg/sm, max 2 mg, D 1)/cycle; Interferon -IFN (3 MU/sm x 3 times/week, x 12 weeks)

SUMMARY:
Rituximab plus CVP and Interferon chemoimmunotherapy for newly diagnosed Follicular Lymphoma with FLIPI index >2

DETAILED DESCRIPTION:
This study is a multicentric trial evaluating the efficacy of the CVP chemotherapy + Interferon (IFN) + Rituximab induction regimen in patients aged 18 to 75 years with newly diagnosed follicular NHL.

Follicular non Hodgkin's lymphoma's (FL), as defined by the REAL Classification, are usually characterized by a slowly progressive clinical course, a transient control by standard chemotherapeutic regimen and a pattern of repeated relapses until ultimately progressive and fatal disease.

Most standard first line treatment for advanced FL consists of alkylating-based (CVP) or anthracycline containing regimens, in association with immunomodulating agents such as interferon alpha or the unconjugated chimeric anti-CD20 antibody (rituximab) to target the CD20 antigen highly expressed on follicular lymphoma cells. This strategies have significantly increased the survival of the patients, but relapses still occur. Thus, the treatment of the patients with FL, requires improvements.

IFN alpha has antiproliferative and immunomodulatory properties. Moreover, it has been described a synergistic effect when IFN is given with chemotherapy. This association has significantly improved progression free survival (PFS) and overall survival (OS). Our prior results with 12 weeks of IFN plus CVP as induction treatment, significantly increased PFS when compared with CVP alone (60% median PFS vs. 24%, p: 0.0004).

We also performed a prospective study to analyze the correlation between the duration of remission and MRD in patients who were treated with CVP+IFN . Ninety four percent of patients had a molecular marker (60% bcl-2 translocation and 34% IgH rearrangement). Molecular response, defined as achieving a negative molecular MRD, was achieved in 76% of patients and it was associated with clinical remission. There was also a significant correlation between the duration of remission and a sustained indetectable MRD Anti-CD20 monoclonal antibody (Rituximab) mediates complement dependent cytotoxicity (CDC), antibody dependent cellular cytotoxicity (ADCC) and apoptosis. Rituximab has also shown to sensitize drug-resistant lymphoma cell lines to killing by cytotoxic drugs.

There are some "in vitro" studies that have tested the effect of Rituximab and IFN combination. It's been described that when IFN is given with Rituximab, it favours the expression of CD20 and therefore increases its cytotoxic effect - . Preliminary phase II studies show an increase in response rate with duration of response going up to 12 months. Moreover, there are two clinical studies that have tested the efficacy and tolerability of Rituximab added to IFN-alpha vi- ix. The Nordic Lymphoma Group showed a significant increase in ORR (up to 94%) by adding 5 weeks of IFN to re-treatment with 4 doses of Rituximab in patients who had achieved only a minimal or partial remission. Most of these patients, maintained their responses for more than 24 months. With a similar trial design, Sacchi et al. showed an ORR of 74% (33% of CR) and a median duration of response of 19 months. The combination was safe and most grade 3-4 adverse events (15%) were hematologic toxicity (leuko-neutropenia and thrombocytopenia).

Thus, we hypothesize that the combination of rituximab, with our standard induction regimen using IFN plus CVP might lead to synergistic / additive induction of apoptosis through different pathways in poor prognostic patients with FL, improving our previous results. We also hypothesize that this combination will be able to achieve higher molecular remissions, determined by real-time PCR of Bcl-2 translocation.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years-75 years
* Pathologically confirmed low grade, Follicular B cell lymphoma (WHO Classification Follicular grades 1 and 2) , Marginal zone lymphoma or Lymphocytic lymphoma (excluding CLL and MCL)
* FLIPI score ≥ 2
* Chemotherapy-naïve patients. Previous radiation therapy is allowed, but should have been limited.
* Adequate hepatic (bilirubin or ALT/AST < 2,5 times UNL) and renal function, except for those directly disease-related
* Performance status grade 0 to 3
* Frozen biopsy material obtained at relapse or disease progression should be available for central pathology review and molecular biology studies
* Patient information and written informed consent

Exclusion Criteria:

* Previous evolutive malignancy within 5 years of study entry
* Prior chemotherapy treatment
* Clinically significant cardiac disease, as defined by history of symptomatic ventricular arrhythmias, congestive heart failure or myocardial infarction within 12 months of study entry
* Known positivity for HIV, VHB or VHC
* Pregnant or lactating women. Women of childbearing potential, and all men, unwilling to take appropriate contraceptive measures during and for at least 12 months after cessation of therapy
* Any uncontrolled serious non malignant condition or infection which would likely compromise the study objectives
* Non controlled thyroid disfunction
* Severe Autoimmune disease
* Patients with history of severe neuropsychiatric disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2006-02; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) with the CVP + IFNalfa + Rituximab treatment | August 2012

SECONDARY OUTCOMES:
Overall response (ORR) and complete response (CR) rates. Overall Survival MRD by RT-PCR assay Toxicity | August 2012

CONTACTS AND LOCATIONS:
Overall Officials: Reyes Arranz-Saez, MD, Principal Investigator — Fundación Leucemia y Linfoma, Spain
Locations (1):
- Hospital Universitario de La Princesa, Madrid, Madrid, Spain